CLINICAL TRIAL: NCT07325890
Title: Research on the Application of Decision Tree in Child Life
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHFudanU1212
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Psychosocial Intervention; Non-Randomized Controlled Trials
Keywords: Child Life
MeSH Terms: interventions — Decision Trees

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Applying decision tree of Child Life for children (Experimental): (1) The decision tree for Child Life was applied to conduct Child Life intervention for the children included in the event. (2) The knowledge level of Child Life Specialists was collected before and after the application. (3) The compliance and pain level of the children included in the event were collected. (4) The working effect of Child Life Specialists was cross-evaluated by two Certified Child Life Specialists.
  Interventions: Other: decision tree for Child Life
- Routine Child Life intervention for children (Active Comparator): (1) Routine Child Life intervention was applied for the children included in the event. (2) The knowledge level of Child Life Specialists was collected before and after the application. (3) The compliance and pain level of the children included in the event were collected. (4) The working effect of Child Life Specialists was cross-evaluated by two Certified Child Life Specialists.
  Interventions: Other: Routine Child Life intervention for children

INTERVENTIONS:
Other: decision tree for Child Life — Four training sessions on decision tree for Child Life were conducted for Child Life Specialists. The training content was produced by the research team based on previous literature and clinical experience. After the training, Child Life Specialists will apply the Child Life decision tree in clinical practice to carry out Child Life intervention.
  Arms: Applying decision tree of Child Life for children
Other: Routine Child Life intervention for children — Child Life Specialists will conduct Child Life intervention for children based on their professional knowledge and clinical experience in clinical practice.
  Arms: Routine Child Life intervention for children

SUMMARY:
The purpose of this study is to understand whether the decision tree for Child Life is effective in improving the professional level and working effect of Child Life Specialists. The main questions it aims to answer are:

1. Does the decision tree for Child Life enhance the professional knowledge level of Child Life Specialists?
2. Has the decision tree for Child Life improved the work effectiveness of Child Life Specialists?
3. Has the application of Child Life decision trees improved children's pain levels and compliance?

Researchers will compare the intervention group and the observation group to see if the decision tree for Child Life can enhance the professional level and work effectiveness of Child Life Specialists.

Participants in the intervention group will:

1. Receive training on the application of decision trees for Child Life.
2. Apply the decision tree for Child Life to carry out intervention in Child Life intervention.
3. Participate in knowledge level tests, work effect evaluations, and record the pain levels and compliance of pediatric patients.

Participants in active comparator will:

1. Conduct Child Life intervention based on one's own experience and professional level.
2. Participate in knowledge level tests, work effect evaluations, and record the pain levels and compliance of pediatric patients.

DETAILED DESCRIPTION:
Psychosocial issues, such as behavioral problems, social interaction disorders and learning difficulties, have become important topics in children's health care. These problems not only affect the immediate recovery of the child patients and increase the risk of complications such as delirium, but may also have a profound negative impact on their long-term development.

The application of decision tree for Child Life can provide clinical workers with effective and feasible intervention strategies, promote the standardization of Child Life practices, thereby reducing the psychological trauma of hospitalization on children and improving the overall quality of care for pediatric patients.

This study adopted a non-randomized controlled study and the intervention was carried out at Fudan University Children's Hospital.

Tools such as the "Questionnaire on Knowledge Level of Child Life Specialists" and the "Questionnaire on Evaluation of Work Effect of Child Life Specialists" were used to evaluate the two groups before and after the training respectively, and children's information of the included cases was collected during the process.

ELIGIBILITY:
Inclusion Criteria:

* Have received training in relevant courses on Child Life.
* Have been engaged in clinical practice of Child Life for at least one year.

Exclusion Criteria:

* Those who are currently on internship, in further education, or not directly involved in clinical treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Clinical anxiety and cooperative behavior manifestations of the child patient | From enrollment to the end of intervention at 2 months
  Before and after each intervention, researchers collected on-site the clinical anxiety and cooperative behavior manifestations of the children included in the intervention plan. The scoring range of this scale is from 0 to 5, with a total of six points. A score of 0 indicates ease, 1 indicates discomfort, 2 indicates tension, 3 indicates reluctance, 4 indicates fear, and 5 indicates loss of control. The higher the score, the more resistant the child is to treatment and the poorer the degree of cooperation. It is generally believed that children with a score of 4 or 5 are unable to cooperate with the treatment.

SECONDARY OUTCOMES:
Questionnaire on Knowledge of Child Life Specialists | From enrollment to the end of training at 2 months
  This questionnaire is derived from the ACLP Child Life Specialists(CLS) Knowledge Question Bank, aiming to assist the CLS system in mastering the psychological support, developmental-appropriate care, and service skills required by the profession. In this study, 25 questions were randomly selected from the total question bank to form an online questionnaire. The total score of the questionnaire is set at 100 points, with 4 points assigned to each question, which is used to test the knowledge level of CLS.
Questionnaire on the Evaluation of the Work Effect of Child Life Specialists | Each intervention ended after enrollment
  The content of this questionnaire is based on the ability evaluation list of Child Life Specialists provided by St. Jude Children's Hospital in the United States. It is based on six dimensions: assessment, games, psychological preparation, procedural support, medical education, and family support. Two CCLS who have been trained and certified by the ACLP system are respectively evaluated for their performance in all modules, professional spirit, and overall practical performance. Provide a summary comment and final rating, which are classified into four categories: poor, average, good, and very good.
Competency Level of Child Life Specialists | From enrollment to the end of training at 2 months
  To comprehensively and objectively assess the ability level of Child Life Specialists(CLS) in clinical practice, the research team, based on Dreyfus' skill acquisition model, divided the professional ability of CLS into four consecutive development stages: novice level, advanced beginner level, competent level and proficient level. Cross-validation through simultaneous evaluation by two CCLS is conducted to truly reflect the professional maturity of CLS in complex clinical contexts.
FACES Pain Scale | From enrollment to the end of intervention at 2 months
  FACES Pain Scale in this study was only conducted in specific clinical situations that might cause pain in the children. Specifically, the children patients will be independently evaluated by two trained researchers to ensure the reliability and accuracy of the scores. During this assessment process, researchers comprehensively judged the degree of pain of the children based on their behavioral responses and verbal expressions, and marked the corresponding scores on the visual analogue scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No